CLINICAL TRIAL: NCT00219258
Title: A Randomized, Double-blind, Multi-centre Study to Evaluate the Fficacy and Safety of Zometa as a Treatment in Patients With Bone Metastases of Any Solid Tumors or Multiple Myeloma
Brief Title: Efficacy and Safety of Zoledronic Acid in Patients With Bone Metastases of Any Solid Tumors or Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446E2301
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Treatment of Bone Metastases
MeSH Terms: interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
Zoledronic acid is a medication that slows the breakdown of bone. This study will assess the efficacy and safety of zoledronic acid in Chinese patients with multiple myeloma or other solid tumors with bone metastases.

ELIGIBILITY:
Inclusion Criteria

* Cancer patients (multiple myeloma or other solid tumors) and confirmed evidence of bone lesions
* Significant bone pain

Exclusion Criteria

* Poor renal function
* Use of other investigational drugs within 30 days of visit 2
* Dental or other surgery to the jaw within 6 weeks of screening, or planned during the 4 week study

Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240
Dates: Start 2005-07

PRIMARY OUTCOMES:
To compare in a randomized fashion the effect of zoledronate and pamidronate 90 mg on pain relief as assessed by pain score after 1-dose treatment in patients with bone pain induced by any solid tumors with bone metastases or Multiple Myeloma

SECONDARY OUTCOMES:
Changes in bone markers (urinary N-telopeptide/creatinine ratio, urinary C-telopeptide/creatinine ratio).

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Beijing, Beijing, China